CLINICAL TRIAL: NCT00092989
Title: A Multicenter, Randomized, Double-Blind Study Comparing the Clinical Effects of Intravenous Montelukast With Placebo in Patients With Acute Asthma
Brief Title: Investigation of Intravenous (IV) Administration of an Approved Drug (MK-0476, Montelukast Sodium) for Acute Asthma (MK-0476-288)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-288; MK-0476-288 (Other: Merck Protocol Number); 2004_027 (Other: Merck Registration Number)
Record Dates: First submitted 2004-09-28; First posted 2004-09-29 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Montelukast 7 mg (Experimental): Participants receive montelukast 7 mg intravenously (IV) until until a decision is made for one of the following: (1) discontinuation from the study, (2) discharge from the study site, or (3) admission to the hospital. All randomized participants will receive systemic corticosteroids (60 mg prednisone OR 50 mg prednisolone) orally immediately after the completion of the study drug administration. In addition, all participants will continue to receive standardized treatment in addition to study drug. Standardized treatment may consist of: (1) β-agonist administration beginning 20 minutes after study drug infusion, and every 20 minutes thereafter, as needed; (2) oxygen therapy; and (3) inhaled ipratropium every 60 minutes as needed.
  Interventions: Drug: montelukast sodium
- Placebo (Placebo Comparator): Participants receive placebo IV until until a decision is made for one of the following: (1) discontinuation from the study, (2) discharge from the study site, or (3) admission to the hospital. All randomized participants will receive systemic corticosteroids (60 mg prednisone OR 50 mg prednisolone) orally immediately after the completion of the study drug administration. In addition, all participants will continue to receive standardized treatment in addition to study drug. Standardized treatment may consist of: (1) β-agonist administration beginning 20 minutes after study drug infusion, and every 20 minutes thereafter, as needed; (2) oxygen therapy; and (3) inhaled ipratropium every 60 minutes as needed.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast sodium — Duration of Treatment: 1 dose
  Other Names: MK-0476; montelukast
  Arms: Montelukast 7 mg
Drug: placebo — Duration of Treatment: 1 dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate improved results of treatment for patients entering an emergency department with asthma attacks when given an investigational IV administration of an approved drug (MK-0476, montelukast sodium) in addition to approved standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with acute asthma

Exclusion Criteria:

* Women of child bearing age
* History of Chronic Obstructive Pulmonary Disease (COPD)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2004-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Improvement in forced expiratory volume in 1 second [FEV1] within the first 60 minutes after administration | within the first 60 minutes after administration

SECONDARY OUTCOMES:
Incidence of treatment failures, amount of additional therapy[short-acting B-agonist] required, rate of FEV1 improvement, safety and tolerability | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Camargo CA Jr, Gurner DM, Smithline HA, Chapela R, Fabbri LM, Green SA, Malice MP, Legrand C, Dass SB, Knorr BA, Reiss TF. A randomized placebo-controlled study of intravenous montelukast for the treatment of acute asthma. J Allergy Clin Immunol. 2010 Feb;125(2):374-80. doi: 10.1016/j.jaci.2009.11.015. PMID 20159247